CLINICAL TRIAL: NCT02124954
Title: A Phase I, Open Label Study to Assess the Effects of TA-8995 on the Pharmacokinetics of Midazolam and Digoxin in Healthy Male Subjects
Brief Title: A Preliminary Drug Drug Interaction Study With TA-8995
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xention Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: TA-8995-05
Record Dates: First submitted 2014-04-17; First posted 2014-04-28 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Pharmacokinetic Interactions
MeSH Terms: interventions — TA-8995; Midazolam; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digoxin with/without TA-8995 (Experimental): Digoxin with/without TA-8995
  Interventions: Drug: TA-8995; Drug: Digoxin
- Midazolam with/without TA-8995 (Experimental): Midazolam with/without TA-8995
  Interventions: Drug: TA-8995; Drug: Midazolam

INTERVENTIONS:
Drug: TA-8995
Drug: Midazolam
  Arms: Midazolam with/without TA-8995
Drug: Digoxin
  Arms: Digoxin with/without TA-8995

SUMMARY:
A study in healthy males to look at how multiple doses of TA-8995 affect blood levels and rate of removal of other drugs, using single doses of digoxin and midazolam as examples, to see if there are any potential drug interactions that might affect patients in future studies. The study will examine whether co-administration of TA-8995 affects the pharmacokinetics of digoxin and midazolam measured by area under the curve (AUC).

ELIGIBILITY:
Inclusion Criteria

* Healthy male subjects

Exclusion Criteria

* Receiving any other drug therapy
* Clinically significant medical history
* Abnormal laboratory results or ECGs

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of TA-8995, midazolam and digoxin | Over 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Brooks, Principal Investigator — Covance
Locations (1):
- Covance, Leeds, United Kingdom